CLINICAL TRIAL: NCT00467870
Title: A Two-Arm, Open-Label, Randomized, Multi-Center Pharmacokinetic and Long-Term Safety Study of Intramuscular Injections of 750 mg and 1000 mg Testosterone Undecanoate in Hypogonadal Men
Brief Title: Long-term Safety Study of Intramuscular Injections of 750 mg and 1000 mg Testosterone Undecanoate in Hypogonadal Men
Acronym: TU
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IP157-001
Record Dates: First submitted 2007-04-27; First posted 2007-05-01 (Estimated); Results first posted 2017-03-07 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Hypogonadism; Primary Hypogonadism; Secondary Hypogonadism
Keywords: investigational; testosterone; testosterone undecanoate; TU; Hypogonadism; primary hypogonadism; secondary hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 750 mg dose of testosterone undecanoate
  Interventions: Drug: Testosterone Undecanoate 750 mg
- 2 (Experimental): 1000 mg dose testosterone undecanoate
  Interventions: Drug: Testosterone Undecanoate 1000 mg

INTERVENTIONS:
Drug: Testosterone Undecanoate 750 mg
  Arms: 1
Drug: Testosterone Undecanoate 1000 mg
  Arms: 2

SUMMARY:
To evaluate the pharmacokinetics of TU 750 mg and TU 1000 mg via multiple measurements of serum total testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Male with primary or secondary hypogonadism at least 18 years of age and for study part C2 weighs ≥143.3 lb (≥65 kg)
* Morning screening serum testosterone concentration <300 ng/dL

Exclusion Criteria:

* American Urological Association (AUA) Symptom Score ≥15 or significant prostatic symptoms
* History of carcinoma, tumors or induration of the prostate or the male mammary gland including suspicion thereof
* Screening serum prostate-specific antigen (PSA) level >4 ng/mL or hyperplasia of the prostate (size >75 cm3 as measured by transrectal ultrasonography)
* Past or present liver tumors or acute or chronic hepatic disease with impairment of liver function; liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST]) exceeding 1.5 times upper limit of normal
* History of deep vein thrombosis in the past 5 years or any history of cerebrovascular accident
* Severe acne
* Hypertension (systolic blood pressure >160 mm Hg and diastolic blood pressure >95 mm Hg) or coronary heart disease not stabilized by therapy as assessed by the investigator
* Insulin-dependent diabetes mellitus or uncontrolled non-insulin-dependent diabetes mellitus; patients with diabetes are excluded if screening glycated hemoglobin (HbA1C) level is >9%
* Use of any sex hormones within 28 days (for injectable testosterone preparations) or 7 days (for oral, gel, patch, etc, testosterone preparations) prior to screening visit and throughout the study (exclusive of administered study drug)
* Use of steroidal anabolic drugs or supplements (eg, dehydroepiandrosterone [DHEA]) by any application method within the 28 days prior to first administration of study drug and throughout the study (exclusive of administrated study drug)
* Medication with substances which might interfere with testosterone metabolism within 28 days before the first administration of study drug
* History of sleep apnea Insulin-dependent diabetes mellitus
* Use of steroidal anabolic drugs or supplements by any application method within the 28-days prior to the first administration of the study drug and throughout the study (exclusive of the administered study drug)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 531 (Actual)
Dates: Start 2006-03; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indevus Pharmaceuticals, Inc., Study Director — Sponsor GmbH
Locations (1):
- Indevus Pharmaceuticals, Inc., Lexington, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 531 subjects who were enrolled, 524 subjects received study treatment (at least 1 injection). The 7 enrolled subjects who did not receive treatment (2 in Part A and 5 in Part C) were excluded from all analyses.
Groups:
- A-TU 750 mg: 750 mg testosterone undecanoate (TU) in 3 mL oily solution, intramuscularly (IM) every 12 weeks for up to 3 years in Part A
- A-TU 1000 mg: 1000 mg TU in 4 mL oily solution, IM every 12 weeks for up to 3 years in Part A
- B-TU 750 mg: 1000 mg TU in 4 mL oily solution, IM at baseline, and then 750 mg TU in 3 mL oily solution at week 8 and again every 10 weeks for up to 23 months in Part B
- B-TU 1000 mg: 1000 mg TU in 4 mL oily solution, IM at baseline, week 8, and then every 12 weeks for up to 24 months in Part B
- C-TU 750 mg: 750 mg TU in 3 mL oily solution, IM at baseline, week 4, and then every 10 weeks for up to 20 months in Part C
- C2-TU 750 mg: 750 mg TU in 3 mL oily solution, IM at baseline, week 4, and then every 10 weeks for up to 12 months in Part C2
Period: Overall Study
Arm/Group | A-TU 750 mg | A-TU 1000 mg | B-TU 750 mg | B-TU 1000 mg | C-TU 750 mg | C2-TU 750 mg
Started | 120 | 117 | 22 | 112 | 130 | 23
Completed | 75 | 74 | 18 | 79 | 93 | 21
Not Completed | 45 | 43 | 4 | 33 | 37 | 2
Not completed — Adverse Event | 13 | 9 | 1 | 15 | 15 | 1
Not completed — Protocol Violation | 2 | 1 | 1 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 14 | 21 | 0 | 9 | 10 | 1
Not completed — Lost to Follow-up | 5 | 3 | 1 | 1 | 3 | 0
Not completed — Subject Non-compliance | 3 | 4 | 0 | 1 | 5 | 0
Not completed — Other/Unknown | 8 | 5 | 1 | 5 | 4 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants who were enrolled and received at least 1 injection
Groups:
- A-TU 750 mg: 750 mg TU in 3 mL oily solution, IM every 12 weeks for up to 3 years in Part A
- Total: Total of all reporting groups
Arm/Group | A-TU 750 mg | A-TU 1000 mg | B-TU 750 mg | B-TU 1000 mg | C-TU 750 mg | C2-TU 750 mg | Total
Number analyzed (Participants) | 120 | 117 | 22 | 112 | 130 | 23 | 524
Age, Customized [Mean (Standard Deviation); unit: years] | 55.0 (10.64) | 55.9 (10.77) | 55.3 (10.40) | 52.9 (10.96) | 54.2 (10.25) | 54.5 (10.63) | 54.4 (10.56)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 120 | 117 | 22 | 112 | 130 | 23 | 524
Race/Ethnicity, Customized [Number; unit: participants]
  White | 101 | 106 | 18 | 92 | 97 | 18 | 432
  Asian | 2 | 0 | 1 | 1 | 0 | 0 | 4
  Black | 11 | 8 | 1 | 15 | 16 | 4 | 55
  Hispanic | 3 | 3 | 2 | 4 | 14 | 1 | 27
  Other | 3 | 0 | 0 | 0 | 3 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting Serum Total Testosterone Average Concentration Criteria for Responder During the 3rd Injection Interval in Part C
Description: Responders were participants with serum total testosterone average concentration (Cavg) between 300 and 1000 ng/dL derived from the 3rd injection intensive pharmacokinetic (IPK) interval.
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: Pharmacokinetic (PK) population includes participants who had a minimum of 4 serum total testosterone concentration values within the 3rd injection interval (13 participants were excluded from analysis)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
percentage of participants | 94.0 [89.7 to 98.3]

2. Primary Outcome: Serum Total Testosterone Average Concentration During the 3rd Injection Interval in Part C
Description: Serum total testosterone Cavg derived from the 3rd injection IPK interval
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: PK population includes participants who had a minimum of 4 serum total testosterone concentration values within the 3rd injection interval (13 participants were excluded from analysis)
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
ng/dL | 494.9373 (141.46351)

3. Primary Outcome: Serum Total Testosterone Maximum Concentration During the 3rd Injection Interval in Part C
Description: Serum total testosterone maximum concentration (Cmax) derived from the 3rd injection IPK interval
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
ng/dL | 890.583 (345.1148)

4. Primary Outcome: Serum Total Testosterone Concentration at the End of the Dosing Interval Following the 3rd Injection in Part C
Description: Serum total testosterone concentration at the end of the dosing interval (Ctrough) derived from the 3rd injection IPK interval
Time Frame: Day 70 post injection at week 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
ng/dL | 323.522 (99.1081)

5. Primary Outcome: Percentage of Participants Meeting Serum Total Testosterone Average Concentration Criteria for Responder During the 4th Injection Interval in Part C
Description: Responders were participants with serum total testosterone Cavg between 300 and 1000 ng/dL derived from the 4th injection IPK interval.
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: Steady-state PK population includes all participants in the PK population with non-missing 4th and 5th injection serum total testosterone concentrations (26 participants were excluded from analysis)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
percentage of participants | 96.2 [92.5 to 99.8]

6. Primary Outcome: Serum Total Testosterone Average Concentration During the 4th Injection Interval in Part C
Description: Serum total testosterone Cavg derived from the 4th injection IPK interval
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
ng/dL | 514.2792 (163.11476)

7. Primary Outcome: Serum Total Testosterone Maximum Concentration During the 4th Injection Interval in Part C
Description: Serum total testosterone Cmax derived from the 4th injection IPK interval
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
ng/dL | 837.648 (412.0692)

8. Primary Outcome: Serum Total Testosterone Concentration at the End of the Dosing Interval Following the 4th Injection in Part C
Description: Serum total testosterone Ctrough derived from the 4th injection IPK interval
Time Frame: Day 70 post injection at week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
ng/dL | 342.800 (106.9180)

9. Primary Outcome: Percentage of Participants Meeting Serum Total Testosterone Maximum Concentration Criteria for Success During the 2nd Injection Interval in Part C2
Description: Success was defined as having ≥85% of participants with Cmax ≤1500 ng/dL, ≤5% of participants with Cmax 1800-2500 ng/dL, and no participants with Cmax >2500 ng/dL.
Time Frame: Days 0, 4, 7, 11, 14, and 70 post injection at week 4
Population: Total patient sample/PK sample includes participants who were enrolled, received injection 2, and had at least 1 post-injection 2 IPK sample (no participants were excluded)
Measure: Number; unit: percentage of participants
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
percentage of participants
  Cmax ≤1500 ng/dL | 95.7
  Cmax 1800-2500 ng/dL | 0
  Cmax >2500 ng/dL | 0

10. Primary Outcome: Serum Total Testosterone Average Concentration During the 2nd Injection Interval in Part C2
Description: Serum total testosterone Cavg derived from the 2nd injection IPK interval
Time Frame: Days 0, 4, 7, 11, 14, and 70 post injection at week 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
ng/dL | 449.6455 (157.00582)

11. Primary Outcome: Serum Total Testosterone Maximum Concentration During the 2nd Injection Interval in Part C2
Description: Serum total testosterone Cmax derived from the 2nd injection IPK interval
Time Frame: Days 0, 4, 7, 11, 14, and 70 post injection at week 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
ng/dL | 689.002 (266.9442)

12. Primary Outcome: Serum Total Testosterone at the End of the Dosing Interval Following the 2nd Injection in Part C2
Description: Serum total testosterone Ctrough derived from the 2nd injection IPK interval
Time Frame: Day 70 post injection at week 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
ng/dL | 317.419 (105.3124)

13. Secondary Outcome: Serum Total Testosterone Maximum Concentration in Part A
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, 70, and 84 post injection at week 1, week 12, week 24, and week 36; and post injection at weeks 48, 60, 72, 84, 96, 108, and 120
Population: Total patient sample includes participants who were enrolled and received at least 1 injection; participants without any IPK sample collections were excluded from this analysis (20 from A-TU 750 mg and 11 from A-TU 1000 mg)
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | A-TU 750 mg | A-TU 1000 mg
Number analyzed (Participants) | 106 | 100
ng/dL | 805.867 (308.5417) | 1023.591 (394.3051)

14. Secondary Outcome: Serum Total Testosterone Maximum Concentration in Part B
Time Frame: Post injection at week 1; post injection at week 8; days 0, 4, 7, 11, 14, 21, 28, 42, 56, 70, and 84 post injection at week 20; and post injection at weeks 32, 44, 56, 68, and 80
Population: Total patient sample includes participants who were enrolled and received at least 1 injection; participants without any IPK sample collections were excluded from this analysis (2 from B-TU 750 mg and 12 from B-TU 1000 mg)
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | B-TU 750 mg | B-TU 1000 mg
Number analyzed (Participants) | 20 | 100
ng/dL | 986.364 (330.4247) | 1047.739 (571.1648)

15. Secondary Outcome: Percentage of Participants Meeting Serum Total Testosterone Maximum Concentration Criteria for Success During the 3rd Injection Interval in Part C
Description: Success is defined as having ≥85% of participants with Cmax ≤1500 ng/dL, ≤5% of participants with Cmax 1800-2500 ng/dL, and no participants with Cmax >2500 ng/dL.
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
percentage of participants
  Cmax ≤1500 ng/dL | 92.3 [87.5 to 97.1]
  Cmax 1800-2500 ng/dL | 0 [0 to 0]
  Cmax >2500 ng/dL | 0 [0 to 0]

16. Secondary Outcome: Percentage of Participants With at Least 1 Serum Total Testosterone Level <300 ng/dL at Any Time During the 3rd Injection Interval in Part C
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
percentage of participants | 51.3 [42.2 to 60.3]

17. Secondary Outcome: Percentage of Participants With Serum Total Testosterone Average Concentration ≥300 ng/dL During the 3rd Injection Interval in Part C
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
percentage of participants | 94.9 [90.9 to 98.9]

18. Secondary Outcome: Time to First Serum Total Testosterone Concentration <300 ng/dL Following the 3rd Injection Interval in Part C
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: PK population includes participants who had a minimum of 4 serum total testosterone concentration values within the 3rd injection interval (13 participants were excluded from analysis); an additional 57 participants who did not have serum total testosterone concentrations <300 ng/dL were also excluded from analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 60
days | 50.2 (17.41)

19. Secondary Outcome: Percentage of Participants With Clinical Success During the 3rd Injection Interval in Part C
Description: Clinical success is defined as having both Cavg and Ctrough between 300 and 1000 ng/dL
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
percentage of participants | 53.8 [44.8 to 62.9]

20. Secondary Outcome: Percentage of Participants With Serum Total Testosterone Maximum Concentration ≤1500, >1500 to <1800, 1800 to 2500, and >2500 ng/dL During the 3rd Injection Interval in Part C
Time Frame: Days 0, 4, 7, 11, 14, 21, 28, 42, 56, and 70 post injection at week 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
percentage of participants
  Cmax ≤1500 ng/dL | 92.3 [87.5 to 97.1]
  Cmax >1500-<1800 ng/dL | 7.7 [2.9 to 12.5]
  Cmax 1800-2500 ng/dL | 0 [0 to 0]
  Cmax >2500 ng/dL | 0 [0 to 0]

21. Secondary Outcome: Percentage of Participants Meeting Serum Total Testosterone Maximum Concentration Criteria for Success During the 4th Injection Interval in Part C
Description: as for outcome 15
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
percentage of participants
  Cmax ≤1500 ng/dL | 92.3 [87.2 to 97.4]
  Cmax 1800-2500 ng/dL | 3.8 [0.2 to 7.5]
  Cmax >2500 ng/dL | 0 [0 to 0]

22. Secondary Outcome: Percentage of Participants With at Least 1 Serum Total Testosterone Level <300 ng/dL at Any Time During the 4th Injection Interval in Part C
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
percentage of participants | 37.5 [28.2 to 46.8]

23. Secondary Outcome: Percentage of Participants With Average Serum Total Testosterone Concentration ≥300 ng/dL During the 4th Injection Interval in Part C
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
percentage of participants | 96.2 [92.5 to 99.8]

24. Secondary Outcome: Time to First Serum Total Testosterone Concentration <300 ng/dL Following the 4th Injection Interval in Part C
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: Steady-state PK population includes all participants in the PK population with non-missing 4th and 5th injection serum total testosterone concentrations (26 participants were excluded from analysis); an additional 57 participants who did not have serum total testosterone concentrations <300 ng/dL were also excluded from analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 39
days | 60.6 (17.51)

25. Secondary Outcome: Percentage of Participants With Clinical Success During the 4th Injection Interval in Part C
Description: Clinical success is defined as having both Cavg and Ctrough between 300 and 1000 ng/dL
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
percentage of participants | 62.5 [53.2 to 71.8]

26. Secondary Outcome: Percentage of Participants With Serum Total Testosterone Maximum Concentration ≤1500, >1500 to <1800, 1800 to 2500, and >2500 ng/dL During the 4th Injection Interval in Part C
Time Frame: Days 0, 4, 7, 11, 42, and 70 post injection at week 24
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 104
percentage of participants
  Cmax ≤1500 ng/dL | 92.3 [87.2 to 97.4]
  Cmax >1500 to <1800 ng/dL | 3.8 [0.2 to 7.5]
  Cmax 1800 to 2500 ng/dL | 3.8 [0.2 to 7.5]
  Cmax >2500 ng/dL | 0 [0 to 0]

27. Secondary Outcome: Percentage of Participants by Collapsed Category for Each Parameter of the Male Patient Global Assessment (M-PGA) at Day 21 of the 3rd Injection Interval in Part C
Description: M-PGA is a 5-item self-report questionnaire to assess perception of change from pretreatment or baseline in hypogonadal symptoms including confidence/self-esteem, sexual performance, moods/behavior, overall feeling of well-being, and satisfaction with study treatment rated on a 7-point scale where items 1-4 were rated as 1 (very much improved), 2 (much improved), 3 (minimally improved), 4 (no change), 5 (minimally worse), 6 (much worse), 7 (very much worse) and item 5 was rated as 1 (very much satisfied), 2 (much satisfied), 3 (minimally satisfied), 4 (neither satisfied nor dissatisfied), 5 (minimally dissatisfied), 6 (much dissatisfied), 7 (very much dissatisfied). Collapsed ratings: Improved=Very much, much, or minimally improved; Worsened=Very much, much, or minimally worse; No change; Satisfied=Very much, much, or minimally satisfied; Not satisfied=Very much, much, or minimally dissatisfied; No opinion (neither satisfied nor dissatisfied).
Time Frame: Day 21 post injection at week 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 117
percentage of participants
  Confidence or Self-Esteem Improved | 82.6 [75.0 to 90.2]
  Confidence or Self-Esteem No Change | 17.4 [0.8 to 34.0]
  Confidence or Self-Esteem Worsened | 0 [0 to 0]
  Satisfaction with Sexual Performance Improved | 80.0 [71.8 to 88.2]
  Satisfaction with Sexual Performance No Change | 17.4 [0.8 to 34.0]
  Satisfaction with Sexual Performance Worsened | 2.6 [0.0 to 20.6]
  General Moods and Behavoir Improved | 80.9 [72.9 to 88.9]
  General Moods and Behavoir No Change | 19.1 [2.7 to 35.6]
  General Moods and Behavoir Worsened | 0 [0 to 0]
  Overal Feeling of Well-Being Improved | 81.7 [73.9 to 89.5]
  Overal Feeling of Well-Being No Change | 18.3 [1.7 to 34.8]
  Overal Feeling of Well-Being Worsened | 0 [0 to 0]
  Satisfaction with Study Treatment Satisfied | 92.2 [87.1 to 97.3]
  Satisfaction with Study Treatment No Opinion | 7.8 [0.0 to 25.4]
  Satisfaction with Study Treatment Not Satisfied | 0 [0 to 0]

28. Secondary Outcome: Change in Body Mass Index From Baseline to Week 24 in Part C
Description: Difference in Body Mass Index (BMI) from baseline to week 24 calculated from weight (kg) divided by height squared (m2)
Time Frame: Baseline, Week 24
Population: PK population includes participants who had a minimum of 4 serum total testosterone concentration values within the 3rd injection interval (13 participants were excluded from analysis); 1 additional participant did not have a measurement at week 24 and was also excluded from analysis
Measure: Mean (Standard Deviation); unit: kg/m2
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 116
kg/m2 | 0.023 (0.9543)

29. Secondary Outcome: Change in Weight From Baseline to Week 24 in Part C
Time Frame: Baseline, Week 24
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | C-TU 750 mg
Number analyzed (Participants) | 116
kg | 0.06 (3.009)

30. Secondary Outcome: Percentage of Participants With at Least 1 Serum Total Testosterone Concentration >1000, >1100, >1250, and <300 or >1000 ng/dL During the 2nd Injection Interval in Part C2
Time Frame: Days 0, 4, 7, 11, 14, and 70 post injection at week 4
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
percentage of participants
  Cmax >1000 ng/dL | 8.7
  Cmax >1100 ng/dL | 4.3
  Cmax >1250 ng/dL | 4.3
  Cmax <300 or >1000 ng/dL | 60.9

31. Secondary Outcome: Serum Dihydrotestosterone Concentrations During the 2nd Injection Interval in Part C2
Time Frame: Days 0, 4, 7, 11, 14, and 70 post injection at week 4
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
pg/mL
  Day 0 (n=23) | 180.33 (111.646)
  Day 4 (n=20) | 301.85 (188.818)
  Day 7 (n=22) | 322.74 (197.018)
  Day 11 (n=22) | 332.92 (210.534)
  Day 14 (n=21) | 324.74 (191.489)
  Day 70 (n=23) | 230.71 (113.578)

32. Secondary Outcome: Serum Total Testosterone Concentrations in Part C2
Time Frame: Screening; day 0; days 0, 4, 7, 11, and 14 post injection at week 4; weeks 14, 24, 34, and 44
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
ng/dL
  Screening (n=22) | 197.629 (75.8138)
  Day 0 (n=23) | 210.363 (81.6797)
  Day 0 at Week 4 (n=23) | 254.669 (112.7259)
  Day 4 post injection at Week 4 (n=20) | 578.419 (304.6675)
  Day 7 post injection at Week 4 (n=22) | 606.484 (266.4847)
  Day 11 post injection at Week 4 (n=22) | 580.614 (244.3727)
  Day 14 post injection at week 4 (n=21) | 545.236 (234.5882)
  Week 14 (n=23) | 317.419 (105.3124)
  Week 24 (n=23) | 316.215 (126.1430)
  Week 34 (n=22) | 374.698 (161.7627)
  Week 44 (n=20) | 375.797 (136.5283)

33. Secondary Outcome: Percentage of Participants With Serum Total Testosterone Concentrations Outside the Normal Range in Part C2
Description: Serum total testosterone concentrations outside the normal range are categorized as <300 ng/dL (below lower limit of normal range) and >1000 ng/dL (above upper limit of normal range)
Time Frame: Screening; day 0; days 0, 4, 7, 11, and 14 post injection at week 4; weeks 14, 24, 34, and 44
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
percentage of participants
  Screening, <300 ng/dL | 100.0
  Screening, >1000 ng/dL | 0
  Day 0, <300 ng/dL | 91.3
  Day 0, >1000 ng/dL | 0
  Day 0 at Week 4, <300 ng/dL | 78.3
  Day 0 at Week 4, >1000 ng/dL | 0
  Day 4 post injection at Week 4, <300 ng/dL | 15.0
  Day 4 post injection at Week 4, >1000 ng/dL | 5.0
  Day 7 post injection at Week 4, <300 ng/dL | 0
  Day 7 post injection at Week 4, >1000 ng/dL | 9.1
  Day 11 post injection at Week 4, <300 ng/dL | 0
  Day 11 post injection at Week 4, >1000 ng/dL | 4.5
  Day 14 post injection at Week 4, <300 ng/dL | 0
  Day 14 post injection at Week 4, >1000 ng/dL | 4.8
  Week 14, <300 ng/dL | 52.2
  Week 14, >1000 ng/dL | 0
  Week 24, <300 ng/dL | 47.8
  Week 24, >1000 ng/dL | 0
  Week 34, <300 ng/dL | 36.4
  Week 34, >1000 ng/dL | 0
  Week 44, <300 ng/dL | 35.0
  Week 44, >1000 ng/dL | 0

34. Secondary Outcome: Trough Assessments of Serum Total Testosterone Concentrations in Part C2
Time Frame: Screening; day 0; and weeks 4, 14, 24, 34, and 44
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
ng/dL
  Screening (n=22) | 197.629 (75.8138)
  Day 0 (n=23) | 210.363 (81.6797)
  Week 4 (n=23) | 254.669 (112.7529)
  Week 14 (n=23) | 317.419 (105.3124)
  Week 24 (n=23) | 316.215 (126.1430)
  Week 34 (n=22) | 374.698 (161.7627)
  Week 44 (n=20) | 375.797 (136.5283)

35. Secondary Outcome: Serum Total Testosterone Maximum Concentration in Part C2
Time Frame: Screening; day 0; days 0, 4, 7, 11, and 14 post injection at week 4; and weeks 14, 24, 34, and 44
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: ng/dL
Arm/Group | C2-TU 750 mg
Number analyzed (Participants) | 23
ng/dL | 711.343 (257.5643)

ADVERSE EVENTS:
Time Frame: Throughout the study (up to 3 years)
Description: Includes all participants who were enrolled and received at least 1 injection, pooled into groups of maximum TU dose received at any time during the study
Groups:
- TU 750 mg: 750 mg TU in 3 mL oily solution, IM at baseline and during the study in Part A, C, or C2 (includes participants from A-750 mg, C-750 mg, and C2-750 mg)
- TU 1000 mg: 1000 mg TU in 4 mL oily solution, IM at any time during the study in Part A or B (includes participants from A-1000 mg, B-750 mg, and B-1000 mg)
Arm/Group | TU 750 mg | TU 1000 mg
Serious Adverse Events (participants affected / at risk) | 38/272 | 37/252
Other Adverse Events (participants affected / at risk) | 131/272 | 120/252
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TU 750 mg (N=272) | TU 1000 mg (N=252)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arrhythmia superventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 3
Hypertrophic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 3 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Abdonimal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Colitis Ischaemic (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Medical device complication (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 2
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Post procedural swelling (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Stab wound (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Spinal ostheoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Convulsion (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 1 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 0 | 2
Gastroenteritis viral (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TU 750 mg (N=272) | TU 1000 mg (N=252)
Sinusitis (Infections and infestations) | 18 | 13
Upper respiratory tract infection (Infections and infestations) | 15 | 15
Nasopharyngitis (Infections and infestations) | 14 | 14
Bronchitis (Infections and infestations) | 12 | 8
Urinary tract infection (Infections and infestations) | 5 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 11
Back Pain (Musculoskeletal and connective tissue disorders) | 13 | 10
Musculoskelatal pain (Musculoskeletal and connective tissue disorders) | 6 | 12
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 9
Prostatic specific antigen increased (Investigations) | 20 | 10
Fatigue (General disorders) | 17 | 8
Injection site pain (General disorders) | 10 | 15
Prostatitis (Reproductive system and breast disorders) | 15 | 13
Erectile dysfunction (Reproductive system and breast disorders) | 4 | 10
Diarrhoae (Gastrointestinal disorders) | 4 | 11
Nausea (Gastrointestinal disorders) | 4 | 8
Insomnia (Psychiatric disorders) | 12 | 12
Depression (Psychiatric disorders) | 8 | 8
Anxiety (Psychiatric disorders) | 5 | 8
Headache (Nervous system disorders) | 6 | 8
Dysuria (Renal and urinary disorders) | 3 | 8
Acne (Skin and subcutaneous tissue disorders) | 9 | 4
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 10 | 4
Hypertension (Vascular disorders) | 16 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other